CLINICAL TRIAL: NCT00458081
Title: A 12-month Multicentre, Randomised, Double-blind, Placebo-controlled Study With Two Parallel Groups to Assess the Effects of Rimonabant 20 mg in Patients With Abdominal Obesity and Microalbuminuria, With Type 2 Diabetes Mellitus or Dyslipidaemia With or Without Other Cardiometabolic Risk Factors.
Brief Title: Evaluation of the Rimonabant Impact on the Regression of Asymptomatic Damage Caused by Cardiovascular Risk Factors
Acronym: RIALTO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision has been taken in light of recent demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIMON_L_01031; EudraCT # : 2006-002951-33
Record Dates: First submitted 2007-04-06; First posted 2007-04-09 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Obesity; Microalbuminuria; Diabetes Mellitus, Type 2; Dyslipidemia
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rimonabant (Experimental)
  Interventions: Drug: Rimonabant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimonabant — 20 mg once per day + slightly reduced calorie diet
  Arms: Rimonabant
Drug: Placebo — placebo once per day + slightly reduced calorie diet
  Arms: Placebo

SUMMARY:
Primary objective:

* To assess the effect on microalbuminuria levels of treatment with rimonabant 20 mg versus a placebo during a 12 month period.

Secondary objectives:

* Percentage of patients in both arms of the study whose levels of microalbuminuria decrease, stabilise, increase towards macroalbuminuria or are unchanged after 12 months of treatment with rimonabant or placebo.
* To assess the effect of treatment with rimonabant 20 mg versus placebo over a 12 month period on:

  * Weight and waist circumference.
  * Glycaemia profile: fasting glycaemia, fasting insulinaemia and HbA1c.
  * Lipid and lipoprotein profile: triglycerides, total cholesterol, HDL-C, LDL-C, apolipoproteins A1 and B.
  * Inflammatory markers
  * Adipocytokines.
  * Blood pressure.
  * Glomerular filtration rate.
* To assess the quality of life by means of questionnaire filled in.
* Safety parameters

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index > 27 kg/m2 and < 40 kg/m2.
* Waist circumference > 102 cm in men and > 88 cm in women.
* Microalbuminuria >= 20 mg/g creatinine and < 300 mg/g creatinine in at least two of three morning urine samples taken on 3 separate days prior to the baseline visit.
* Type 2 diabetes and/or dyslipidaemia.

Exclusion Criteria:

* Breastfeeding or pregnant women or who expect to become pregnant.
* Non-use of approved methods of contraception in women of child-bearing potential.
* History of very low calorie diet in the 3 months prior to the screening visit (<1200 kcal/day).
* Change in weight > 5 kg in the 3 months prior to the screening visit.
* History of surgery for weight loss (such as vertical banded gastroplasty, gastric by-pass, etc.)
* History of bulimia or anorexia nervosa according to DSM-IV definition.
* Any clinically significant endocrine disorder, in the opinion of the investigator, especially known alterations in the blood concentration of TSH and free T4.
* Type 1 Diabetes
* Triglyceridaemia > 400 mg/dl (4.52 mmol/l)
* Severe renal dysfunction
* Chronic Hepatitis or clinically known significant liver disease or ALT and/or AST > 3x the upper limit of the normal range at the screening visit.
* Hypertension at the screening visit.
* Presence of any condition (medical, including clinically significant abnormal laboratory tests, physiological, social or geographical) actual or anticipated that the investigator feels would compromise the patient's safety or limit his/her successful participation to the study.
* History of abuse of alcohol or other substances (except smoking).
* Hypersensitivity or intolerance to the active ingredient or any of the excipients, such as lactose.

Concomitant medication prior to the screening visit

* Administration of any treatment undergoing clinical investigation (drug or medical device) in the 30 days prior to the screening visit.
* Previous treatment with rimonabant.
* Administration of any of the following products in the 3 months prior to the screening visit

  * Anti-obesity drugs (such as, sibutramine or orlistat).
  * Other weight loss drugs (phentermine,amphetamines).
  * Weight loss herbal preparations.
  * Nicotinic acid, fibrates, bile acid sequestrants or Omega 3 drugs (e.g. Omacor).
  * Prolonged use (more than a week) of systemic corticosteroids or neuroleptics
  * Antidepressants (including bupropion)
  * Insulin, thiazolidinediones, α-glucosidase inhibitors, meglitinides or any group of antidiabetic drugs (except combination of biguanides and sulfonylureas)
* In type 2 diabetes patients, start of or change in treatment with sulfonylureas and/or metformin, in the 4 weeks prior to the screening visit.
* Start of or change in treatment with antihypertensive drugs in the 12 weeks prior to the screening visit.
* Start of or change in treatment with statins and/or ezetimibe in the 8 weeks prior to the screening visit.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2007-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Relative change in the microalbuminuria level. | between baseline visit and Month 12

SECONDARY OUTCOMES:
Percentage of patients whose albuminuria levels decrease, stabilise, are progressing towards macroalbuminuria, are unaltered. | between baseline visit and Month 12
Relative change and absolute change of Weight, Waist circumference, Body mass index (weight and height), Specific lipid parameters, Glycaemia control parameters, Proinflammatory markers, Adipocytokines, Glomerular filtration rate, Blood pressure | between baseline visit and Month 12
Evaluation of the Quality of Life (questionnaire IWQOL). | at baseline visit and at 3, 6 and 12 months visit
Safety (including neuropsychiatric events) and Laboratory assessments. | at each visit and at baseline, 3, 6 and 12 month visits

CONTACTS AND LOCATIONS:
Overall Officials: José Mª Taboada, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Barcelona, Spain